CLINICAL TRIAL: NCT00003273
Title: Dose Intensive Chemotherapy for Children Less Than Ten Years of Age Newly-Diagnosed With Malignant Brain Tumors: A Pilot Study of Two Alternative Intensive Induction Chemotherapy Regimens, Followed by Consolidation With Myeloablative Chemotherapy (Thiotepa, Etoposide and Carboplatin) and Autologous Stem Cell Rescue
Brief Title: Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Children With Newly Diagnosed Brain Tumor
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066174; NYU-P9712; NCI-V98-1400
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma; Retinoblastoma; Sarcoma
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; extraocular retinoblastoma; childhood choroid plexus tumor; localized unresectable neuroblastoma; previously untreated childhood rhabdomyosarcoma; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood medulloblastoma; newly diagnosed childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Retinoblastoma; Sarcoma; Choroid Plexus Neoplasms | interventions — Filgrastim; Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Leucovorin; Methotrexate; Temozolomide; Thiotepa; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: leucovorin calcium
Drug: methotrexate
Drug: temozolomide
Drug: thiotepa
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of different regimens of combination chemotherapy followed by peripheral stem cell transplantation in treating children who have newly diagnosed brain tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Investigate the toxicity of and response rate to an intensification of an induction chemotherapy regimen (regimen A: cisplatin, vincristine, cyclophosphamide, and etoposide) by incorporation of high-dose methotrexate with leucovorin calcium rescue in patients with primitive neuroectodermal tumors and evidence of leptomeningeal dissemination (M1, M2, or M3).
* Investigate the toxicity of and response rate to a new dose intensive induction chemotherapy regimen (regimen C: vincristine, carboplatin, and temozolomide) in children under ten years of age who are newly diagnosed with either high grade gliomas or diffuse intrinsic pontine tumors. (Regimen B closed to accrual effective 3/30/2000; regimen C open to accrual effective 7/21/2000)
* Investigate the feasibility of utilizing regimen C chemotherapy followed by consolidation with myeloablative chemotherapy and autologous stem cell (either bone marrow and/or peripheral blood) rescue in these patients. (Regimen B closed to accrual effective 3/30/2000; regimen C open to accrual effective 7/21/2000)
* Investigate the toxicity of and response rate to an intensification of induction regimen A chemotherapy by incorporation of high-dose methotrexate with leucovorin calcium rescue in patients with primitive neuroectodermal tumors and evidence of leptomeningeal dissemination (M1, M2, or M3).
* Estimate the time to disease progression and the pattern of relapse in patients who do not have radiographic or cytologic evidence of residual disease at the time of consolidation chemotherapy and who, therefore, do not receive post consolidation irradiation.
* Estimate the time to disease progression and the pattern of relapse in patients who have radiographic or cytologic evidence of residual disease at the time of consolidation chemotherapy and who, therefore, receive post consolidation irradiation.
* Assess the morbidity and mortality of the consolidation chemotherapy regimen following either regimen C or the intensified regimen A in these patients. (Regimen B closed to accrual effective 3/30/2000; regimen C open to accrual effective 7/21/2000)
* Assess the impact that irradiation avoidance or the administration of reduced volume craniospinal and/or focused field local irradiation has on neuropsychometric, endocrinological functions, and physical growth.

OUTLINE: This is a two regimen study based on disease characteristics.

Patients in regimens A, B, and C undergo leukapheresis after receiving filgrastim (G-CSF) by subcutaneous (SC) injections.

* Regimen A: Patients without evidence of neuraxis dissemination receive five 21 day courses of the following chemotherapy: cisplatin IV over 6 hours on day 0; etoposide and cyclophosphamide IV over 1 hour on days 1 and 2; vincristine IV on days 0, 7, and 14 of courses 1, 2, and 3; and G-CSF SC beginning on day 3 of each course and continuing until blood counts recover or up to 48 hours before the start of the next course. Patients with evidence of neuraxis dissemination also receive high-dose methotrexate IV over 4 hours on day 3 and leucovorin calcium orally or by IV bolus starting 24 hours prior to methotrexate and continuing every 6 hours until methotrexate levels have diminished.
* Regimen B (closed to accrual effective 3/30/2000): Patients receive three 21-28 day courses of the following chemotherapy: vincristine IV on days 0, 7, and 14 of each course; carboplatin IV over 4 hours on days 3 and 4 of each course; oral procarbazine daily on days 0-4; oral lomustine on days 3 and 4; and G-CSF SC daily beginning 24 hours following the last dose of carboplatin and continuing until blood counts recover or up to 48 hours before the start of the next course. On day 7 of each course, patients also receive peripheral blood stem cell (PBSC) reinfusion following chemotherapy. Oral lomustine is administered only for the first two courses.
* Regimen C (open to accrual effective 07/21/2000): Patients receive four 28 day courses of the following chemotherapy: carboplatin IV over 4 hours on days 0 and 1 of each course; vincristine IV on days 0, 7, and 14 of the first three courses only; oral temozolomide daily on days 0-4; and G-CSF SC daily beginning on day 5 and continuing until blood counts recover.

After regimen A, B, or C and in the absence of disease progression, patients undergo consolidation myeloablative chemotherapy by receiving carboplatin IV over 4 hours on days -8, -7, and -6, and then thiotepa IV over 3 hours followed by etoposide IV on days -5, -4, and -3. Patients with malignant gliomas or unbiopsied diffuse intrinsic pontine tumors do not receive etoposide. On day 0, patients are reinfused with autologous PBSC. Following recovery from consolidation chemotherapy, patients with radiographic or cytologic evidence of residual disease undergo radiotherapy.

Patients are followed at 3 months, then every 3 months for the first 2 years, then every 6 months for years 2-4, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 96 patients (73 for regimen A and 23 for regimen C) will be accrued for this study. (Regimen B closed to accrual effective 3/30/2000.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant, newly diagnosed brain tumor

Regimen A:

* Posterior fossa medulloblastoma/primitive neuroectodermal tumor (PNET):

  * All stages, under 3 years at diagnosis OR
  * High stage (local residual tumor postoperatively and/or neuraxis or extraneural dissemination), 3-10 years at diagnosis
* Supratentorial PNET, pineoblastoma, cerebral neuroblastoma, ependymoblastoma, medulloepithelioma, medullomyoblastoma:

  * All stages, under 10 years at diagnosis
* Brainstem PNET:

  * All stages, irrespective of extent of resection, under 10 years at diagnosis
* Ependymoma or anaplastic ependymoma:

  * All stages, any location (except primary spinal cord ependymoma), under 3 years at diagnosis OR
  * Local residual tumor postoperatively and/or neuraxis dissemination, any location, 3-10 years at diagnosis
* Supratentorial ependymoma:

  * All stages, irrespective of extent of resection, under 10 years at diagnosis, excluding gross totally resected (confirmed by postoperative MRI) low grade ependymoma not invading the ventricular system
* Metastatic retinoblastoma:

  * Previously untreated (except for cryosurgery or laser surgery), under 10 years at presentation of metastatic disease
* Primary atypical teratoid/rhabdoid tumors of the CNS:

  * Under 10 years at diagnosis
* Choroid plexus carcinoma:

  * Incompletely resected, all sites, under 10 years at diagnosis

Regimen C:

* Anaplastic astrocytoma, glioblastoma multiforme, anaplastic oligodendroglioma, anaplastic ganglioglioma, other anaplastic mixed gliomas:

  * Under 10 years at diagnosis
* Diffuse intrinsic pontine tumors:

  * Unbiopsied, under 10 years at diagnosis

The following diagnoses are not eligible:

* Myxopapillary ependymoma of the spinal cord, low grade brainstem astrocytoma, primary CNS lymphoma or solid leukemic lesion (i.e., chloroma, granulocytic sarcoma), or primary CNS germ cell tumor

PATIENT CHARACTERISTICS:

Age:

* Under 10 at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGPT less than 2.5 times upper limit of normal

Renal:

* Creatinine clearance greater than 60 mL/min

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior corticosteroids allowed
* No concurrent corticosteroids for the sole purpose of antiemesis

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 1997-11

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L. Finlay, MB, ChB, Study Chair — NYU Langone Health
Locations (19):
- United States (17):
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Maine Children's Cancer Program, Scarborough, Maine
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital of Omaha, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Beth Israel Hospital North, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Children's Hospital, Buenos Aires, Buenos Aires, Argentina
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada